CLINICAL TRIAL: NCT00644098
Title: The Effect and Dose-response of Soluble Fibre Blend and Medium Chain Triglycerides (MCT) on Body Composition and Cardiometabolic Risk Factors in Overweight and Obese Adults: a Double-blind, Placebo-controlled Study.
Brief Title: Effect of a Soluble Fibre Blend and Medium Chain Triglycerides on Body Composition and Cardiometabolic Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Center for Functional Medicine (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: People Who Are Overweight or Obesity
MeSH Terms: conditions — Obesity | interventions — Cellulose; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): cellulose and soybean oil
  Interventions: Dietary Supplement: cellulose and soybean oil
- Intervention (Experimental): soluble fibre complex and medium chain triglycerides
  Interventions: Dietary Supplement: soluble fibre complex and medium chain triglycerides

INTERVENTIONS:
Dietary Supplement: soluble fibre complex and medium chain triglycerides
  Arms: Intervention
Dietary Supplement: cellulose and soybean oil
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether the addition of capsules containing soluble fibre complex emulsified with medium chain triglycerides and taken before with meals will lead to a significant amount of weight loss, reduced glycemic volatility and diminished cardio metabolic risk factors in overweight and obese individuals when compared to a placebo control.

We believe that those participants taking 3-6 capsules per day of the treatment capsules over a 14 week period will loose a significant amount of weight compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27 - 35 kg/m2

Exclusion Criteria:

-

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
weight loss | baseline, biweekly and final visit

SECONDARY OUTCOMES:
glycemic volatility and cardio metabolic risk factors | baseline and final visit

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Durance, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Canadian Center for Functional Medicine, Coquitlam, British Columbia, Canada